CLINICAL TRIAL: NCT04281849
Title: Pilot Study of a Moderate- to High-Intensity Home-based Rehabilitation Program in Older Adults Hospitalized for Heart Failure: The Balance, Aerobic Capacity, Mobility and Strength (BAMS-HF) Program.
Brief Title: Balance, Aerobic Capacity, Mobility and Strength in Patients Hospitalized for Heart Failure (BAMS-HF) Program
Acronym: BAMS-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kelsey Flint, Staff Cardiologist, VA Eastern Colorado Health Care System
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-1783; 1R03AG064371-01 (NIH)
Record Dates: First submitted 2020-02-17; First posted 2020-02-24 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure; Heart Failure With Preserved Ejection Fraction; Heart Failure, Systolic; Heart Failure, Diastolic; Heart Failure，Congestive; Heart Failure; With Decompensation; Heart Failure Acute; Heart Failure With Reduced Ejection Fraction
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic; Heart Failure, Diastolic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Patients in the usual care arm will receive educational material from the Heart Failure Society of America (HFSA) with the current recommendations for exercise for patients with heart failure.
- BAMS-HF Program (Experimental)
  Interventions: Behavioral: BAMS-HF Program

INTERVENTIONS:
Behavioral: BAMS-HF Program — BAMS-HF Program (intervention) arm will consist of 3 in-home sessions (45-60 min ea) per week for 12 weeks with the study physical therapist. The study physical therapist will transition appropriate participants to virtual in-home visits (i.e. telerehabilitation) for some visits. The study physical therapist will design individualized exercise programs first targeting strength, then mobility and balance, and finally, aerobic capacity. Exercises will be progressive, with the goal of an 8 repetition maximum for each strength component, 80% completion rate for balance/mobility components and targeting a moderate rate of perceived exertion for aerobic components.
  Interviews: There will be a recorded interview after the last session of the study to get participants' opinion of the program, suggestions for improvement and description of any barriers to participating in the program fully.
  Arms: BAMS-HF Program

SUMMARY:
This is a pilot randomized trial of the BAMS-HF (Balance, Aerobic capacity, Mobility and Strength in patients hospitalized for Heart Failure) Program versus usual care. The BAMS-HF Program pilot study is an initial step in eventually creating a comprehensive, patient-centered, primarily home-based rehabilitation intervention aimed at preventing worsening disability and dependence among older adults hospitalized for HF. The BAMS-HF Program will enroll patients hospitalized for HF (or with HF as an active problem during hospitalization) within the past 4 weeks and will engage patients during the vulnerable post-discharged period. The objective of this pilot study is to test the feasibility, acceptability and preliminary effect of the BAMS-HF Program in older (>/= 65 years) adults hospitalized for HF. The BAMS-HF Program will begin within 4 week of hospital discharge and be administered 3 times weekly for 12 weeks in the patient's home upon discharge. Patients who are able to safely complete the program without in-person assistance will transition to telehealth (aka telerehabilitation) visits. The BAMS-HF Program is innovative because it is home-based, and will utilize rigorous, progressive exercises across multiple domains of physical function. The estimated preliminary effect size will be measured with the Short Physical Performance Battery (SPPB), a well-validated measure that predicts incident mobility/disability and falls in the geriatric population.

Aim #1: To assess the feasibility of the BAMS-HF Program by measuring 1) study enrollment rate, 2) proportion of prescribed sessions that were actually performed, 3) proportion of patients completing full baseline assessment and outcome measures

Aim #2: To assess the acceptability of the BAMS-HF Program with qualitative interviews of participants in the intervention arm that will ask about their experience in the program, any aspects of the intervention they recommend changing and whether patients would recommend the program to others. Reason for declining or stopping participation in the study will also be recorded and considered in adjusting the study protocol.

Aim #3: To estimate the preliminary intervention effect by investigating the difference in change in SPPB between the BAMS-HF Program arm and the usual care arm.

ELIGIBILITY:
Inclusion Criteria:

* 55 years old or older
* Hospitalized for HF or with HF as an active problem during hospitalization
* SPPB >/=10

Exclusion Criteria:

* Irreversible orthopedic or neurologic disease that severely limits mobility
* Active cancer diagnosis except non-melanoma skin cancer
* Dementia
* Life expectancy of < 6 months
* Uncontrolled/untreated ventricular tachycardia or ventricular fibrillation
* Advanced heart failure with expectation of left ventricular assist device or transplant in the next 6 months
* Any major surgery in the past 30 days or planned in the next 10 weeks
* Discharge to a skilled nursing facility and/or home with home healthcare physical therapy (home health care nurse or occupational therapist is ok)

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruiting patients into the study | Monthly, up to 30 months
  Number of patients enrolled in the study each month
Acceptability of the intervention to patients randomized to the intervention arm | At the end of the intervention period for each patient (week 12 or at time of study dropout)
  Qualitative interviews of participants in the intervention arm will ask about their experience in the program, any aspects of the intervention they recommend changing and whether patients would recommend the program to others. Reason for declining or stopping participation in the study will also be recorded and considered in adjusting the study protocol.
Feasibility of the protocol for patients randomized to the intervention arm | At the end of the intervention period for each patient (week 12 or at time of study dropout)
  Proportion of prescribed sessions that were actually performed

SECONDARY OUTCOMES:
Change in Short Physical Performance Battery, which is scored from 0-16, with higher numbers indicating better functional status | At the end of 12 weeks of study enrollment for each patient
  Estimate the preliminary effect of the BAMS-HF Program on change in the Short Physical Performance Battery from baseline to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No